CLINICAL TRIAL: NCT06323460
Title: A Pilot Study of Adaptive De-Intensified Radiotherapy Using Circulating Tumor DNA in HPV- Associated Oropharyngeal Cancer
Brief Title: Adaptive De-intensified Radiotherapy Using Circulating Tumor DNA in HPV- Associated Oropharyngeal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sujith Baliga, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23083; NCI-2024-00904 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Specimen Handling; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Congresses as Topic; Radiation; Paclitaxel; Taxes; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (reduced > 95% of TTMV, external beam radiotherapy) (Experimental): Patients undergo external beam radiotherapy daily for 5 days a week for 4 weeks. Patients also receive cisplatin IV weekly or every 3 weeks or carboplatin/paclitaxel IV weekly at the discretion of treating physician for 4 weeks. Patients undergo blood sample collection for circulating tumor DNA testing at week 4.
  Patients with reduced > 95% of TTMV undergo external beam radiotherapy QD 5 days a week for 5 weeks. Patients also receive cisplatin IV weekly or every 3 weeks or carboplatin/paclitaxel IV weekly at the discretion of treating physician for 5 weeks. Patients also undergo blood sample collection during screening and throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Arm II (not reduced > 95% of TTMV, external beam radiotherapy) (Active Comparator): Patients undergo external beam radiotherapy daily for 5 days a week for 4 weeks. Patients also receive cisplatin IV weekly or every 3 weeks or carboplatin/paclitaxel IV weekly at the discretion of treating physician for 4 weeks. Patients undergo blood sample collection for circulating tumor DNA testing at week 4.
  Patients without reduced > 95% of TTMV undergo external beam radiotherapy daily for 5 days a week for 7 weeks. Patients also receive cisplatin IV weekly or every 3 weeks or carboplatin/paclitaxel IV weekly at the discretion of treating physician for 7 weeks. . Patients also undergo blood sample collection during screening and throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Radiation: External Beam Radiation Therapy — Undergo external beam radiotherapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well using circulating tumor deoxyribonucleic acid (DNA) to guide lower dose radiation therapy works in treating patients with human papillomavirus infection (HPV)-associated oropharyngeal cancer. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Recently, a blood test has been developed to detect the human papillomavirus in the blood and determine how many viral particles are present. Researchers want to compare any good and bad effects of using the lower dose radiation therapy with chemotherapy compared to the usual standard of care dose chemotherapy in patients who clear the human papillomavirus particles from their blood.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the 3-month post-treatment positron emission tomography (PET) response rate in patients who have a favorable tumor tissue modified viral (TTMV) tumor profile (defined as >= 200 copies/mL and reduced to > 95% of this value by week 4).

SECONDARY OBJECTIVES:

I. To assess 2-year progression free survival and toxicity in the reduced dose chemo-radiation arm.

II. To determine acute and late toxicity as measured by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v 5.0).

III. To compare changes in the MD Anderson Dysphagia Inventory (MDADI) of reduced dose radiation to the current standard of care (69.96 Gy).

IV. To determine whether integration of HPV into the host genome is associated with circulating TTMV clearance profiles during chemoradiation (CRT).

OUTLINE:

Patients undergo external beam radiotherapy daily for 5 days a week for 4 weeks. Patients also receive cisplatin intravenously (IV) weekly or every 3 weeks or carboplatin/paclitaxel IV weekly at the discretion of treating physician for 4 weeks. Patients undergo blood sample collection for circulating tumor DNA testing at week 4, and then are assigned to 1 of 2 arms based on the results.

ARM I: Patients with reduced > 95% of TTMV undergo external beam radiotherapy once daily (QD)5 days a week for 5 weeks. Patients also receive cisplatin IV weekly or every 3 weeks or carboplatin/paclitaxel IV weekly at the discretion of treating physician for 5 weeks. Patients undergo PET/computed tomography (CT) scan throughout the trial. Patients also undergo blood sample collection during screening and throughout the trial.

ARM II: Patients without reduced > 95% of TTMV undergo external beam radiotherapy daily for 5 days a week for 7 weeks. Patients also receive cisplatin IV weekly or every 3 weeks or carboplatin/paclitaxel IV weekly at the discretion of treating physician for 7 weeks. Patients undergo PET/CT scan throughout the trial. Patients also undergo blood sample collection during screening and throughout the trial.

After completion of study treatment, patients are followed every 3 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of squamous cell carcinoma of the oropharynx (unknown primary, base of tongue, tonsil, oropharyngeal walls, soft palate). Cytologic or fine needle aspiration (FNA) confirmation is sufficient if a biopsy of the primary tumor is not feasible
* P16 positive immunohistochemical staining. FNA may be used as the sole diagnostic tissue. If staining was done at an outside hospital, central review by the Ohio State University (OSU) department of pathology must occur prior to trial enrollment
* Clinical stage T0, N1-N2, T1-2, N1-N2, T3-T4, N0-2 (American Joint Committee on Cancer [AJCC] 8th edition) including no evidence of distant metastases based on general history, imaging, physical examination, and examination with laryngopharyngoscopy
* Clinical or radiographic evidence of measurable disease at the primary site or lymph nodes. Simple tonsillectomy or excision of primary without removal of nodal disease is permitted, as is excision of gross nodes but with intact primary site
* Fludeoxyglucose F-18 (FDG) PET/CT from the base of skull to the mid-thigh is mandatory and patients cannot be enrolled without a pretreatment PET/CT. PET/CT must be completed prior to enrollment
* Pretreatment tumor tissue modified HPV virus (TTMV-HPV) particles present in plasma cell free DNA value of >= 200 copies/mL at baseline
* Patients must provide their smoking history prior to enrollment. Patients must have =< 10 pack years of smoking. The number of pack years will be calculated using the following formula: Frequency of smoking (cigarettes/day) x duration of cigarette smoking (years)/20
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Age >= 18
* Absolute neutrophil count: ≥ 1500/mcL (within 14 days prior to registration)
* Platelets: >= 100,000/mcL (within 14 days prior to registration)
* Hemoglobin >= 8.0 g/dL (use of transfusion or other intervention to achieve this is acceptable) (within 14 days prior to registration)
* Total bilirubin >= 1.5 x institutional upper limit of normal (within 14 days prior to registration)
* Aspartate transaminase (AST) or alanine transaminase (ALT) >= 3.0 x institutional upper limit of normal (within 14 days prior to registration)
* Serum creatinine =< 1.5 x institutional upper limit of normal or creatinine clearance >= 50 mL/min (Cockcroft-Gault Formula) (within 14 days prior to registration)
* Human immunodeficiency virus (HIV) infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible
* Patients with known positive hepatitis B surface antigen indicating acute or chronic infection would make patient ineligible unless viral load becomes undetectable on suppressive therapy
* Patients with history of hepatitis C virus must have been treated and cured
* For women of childbearing potential, negative serum or urine pregnancy test within 14 days of registration
* Patient or legally authorized representative must provide study specific informed consent prior to study entry

Exclusion Criteria:

* Recurrent disease
* Clinical or radiographic evidence of metastatic disease or adenopathy below the clavicles
* Cancers from an oral cavity site, even if p16 positive
* Patients with simultaneous primary cancers or separate bilateral primary tumors will be excluded, except for patients with bilateral tonsil cancers
* Prior invasive malignancy (except non-melanoma skin cancer) unless disease free for a minimum of 3 years
* Prior systemic chemotherapy or immunotherapy
* Prior radiotherapy that would result in overlap of radiation fields
* Severe active co-morbidity defined as: Unstable angina or congestive heart failure requiring hospitalization in the last 6 months. Condition requiring systemic treatment with steroids or immunosuppressive medications within 14 days of registration
* Patients with active autoimmune disease requiring systemic treatment (disease modifying agents, corticosteroids, or immunosuppressive drugs
* Patients who are pregnant, nursing, or expected to conceive or father children
* Patients who are allergic to cisplatin, carboplatin, or paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Positron emission tomography complete response | At 3 months
  Will be evaluated using the Hopkins Criteria which predicts Overall Survival (OS) and Progression-free survival (PFS) in patients with HPV positive oropharyngeal cancers. Separate scores are given for the primary tumor, right neck, and left neck. The activity in the internal jugular vein (IJV) is taken as background blood pool for reference. A score of 1 is consistent with a complete metabolic response, a score of 2 is associated with likely complete metabolic response, a score of 3 is likely inflammatory changes, and a score of 4 is considered likely residual tumor. The overall assessment is denoted by the overall score, which is the highest score among the scores for the primary tumor and right and left neck.

SECONDARY OUTCOMES:
Progression free survival | At 2 years
  Will be will be analyzed using Kaplan Meier methods.
Incidence of adverse events | Up to 1 year
  The treating physician will evaluate all adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Any adverse event which changes CTCAE grade over the course of a given episode will have each change of grade recorded in the electronic medical record.
Quality of life (QOL) | Up to 1 year
  Will be measured by the MD Anderson Dysphagia Inventory (MDADI) global QOL score. The MDADI is a 20-item self-administered patient reported dysphagia assessment instrument and incorporates global, functional, emotion, and physical subscales. Two overall scores are obtained which include the global and composite scores. The global score is from a single item and the composite score summarizes the remaining 19 items as a weighted average of the physical, emotional, and functional subscales. The scores range from 0 (extremely low functioning) to 100 (high functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Sujith Baliga, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu